CLINICAL TRIAL: NCT07376486
Title: Duodenal Recellularization Via Electroporation Therapy as an Early Treatment for Type 2 Diabetes Mellitus (DREAM-1 Study)
Brief Title: Duodenal ReCET as an Early Treatment for Type 2 DM
Acronym: DREAM-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Stephen KK Ng, Principal Investigator, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2025.801
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabete Mellitus; T2 Diabetes and Fatty Liver Disease (Non-alcoholic Origin)
MeSH Terms: conditions — Diabetes Mellitus; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Endoscopic duodenal recellularization via electroporation therapy (ReCET) (Experimental): ReCET procedure entails the ablation of the duodenal mucosa with irreversible electroporation (IRE)
  Interventions: Procedure: ReCET treatment

INTERVENTIONS:
Procedure: ReCET treatment — The ReCET procedure utilizes the ReCET catheter to deliver non-thermal pulsed electric field to the duodenum to induce cell regeneration. The catheter is introduced to the duodenum through the mouth using a guide wire and the therapy is applied to treat the duodenum under endoscopic visualisation, starting from D4 and repeated proximally. Approximately 10-18 cm of axial length of the duodenum is treated.

SUMMARY:
This study is designed to evaluate the efficacy and safety of endoscopic duodenal re-cellularization therapy in individuals with in patients with a recent diagnosis of type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This is a prospective, single-armed, feasibility study enrolling individuals with a recent diagnosis of type 2 diabetes. Participants will be followed for 6 months for the primary endpoint and 2 years in total.

ELIGIBILITY:
Inclusion Criteria:

* Duration of T2DM </= 2 years
* HbA1c </= 7.5%
* On 0-1 oral diabetes medications

Exclusion Criteria:

* Previous treatment with ReCET or similar procedure
* Previous GI surgery that could preclude the ability to perform ReCET, or acute gastric and duodenal pathology that increased the risk of ReCET
* Type I DM, DM secondary to specific disease or having any history of ketoacidosis
* Fasting C-peptide level <0.5ug/L
* Any inflammatory disease of the gastrointestinal tract such as Crohn's disease
* Abnormal pathologies or conditions of the gastrointestinal tract, including duodenal polyps, ulcers or upper gastrointestinal bleeding conditions within 3 months of study
* Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/microliter or known coagulopathy
* Currently taking prescription antithrombotic therapy (e.g., anticoagulant or antiplatelet agent) within 10 days prior to study and/or there is a need or expected need to use during the study period
* Currently taking medications known to cause significant weight gain or weight loss (e.g. chemotherapeutics)
* Patients who have used non-steroidal analgesics and anti-inflammatory drugs (NSAID) and corticosteroids in the past 1 month
* Underlying uncontrolled endocrine problem that leads to obesity, including and not limited to hypothyroidism, Cushing syndrome and eating disorder.
* Patients with contra-indications to endoscopy
* Malignancy
* Diagnosis of autoimmune connective tissue disorder (e.g. lupus erythematosus, scleroderma)
* Pregnant or breast feeding
* ASA grade IV & V
* Mental or psychiatric disorder; Drug or alcohol addiction
* Other cases deemed by the examining physician as unsuitable for safe treatment
* Refusal to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-08-30 (Estimated); Study Completion 2032-02-28 (Estimated)

PRIMARY OUTCOMES:
HbA1c ≤6.5% without glucose lowering drugs | 6 months post-procedure
  Proportion of participants with HbA1c ≤6.5% without glucose lowering drugs

SECONDARY OUTCOMES:
HbA1c | 24 months post-procedure
  Change in HbA1c (%) from baseline to Month 24
Total body weight loss (%TBWL) | 24 months post-procedure
  Percent total body weight loss (%TBWL) from baseline to Month 24
Incidence of adverse events | within 30 days post-procedure
  Adverse events relating to endoscopic intervention, graded according to the Common Terminology Criteria for Adverse Events (CTCAE)
Body fat percentage | 24 months post-procedure
  Changes in body fat percentage - measured by bioelectrical impedance analysis from baseline to Month 24
Change in Quality of Life | 24 months post-procedure
  measured by 36-Item Short Form Survey (SF-36) questionnaire - (score 0:worst - 100:best) from baseline to Month 24
Hepatic steatosis index | 24 months post-procedure
  level from baseline to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ng, FRCSEd(Gen), Principal Investigator — Prince of Wales Hospital, the Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided